CLINICAL TRIAL: NCT04826640
Title: A Prospective Observational Study to Evaluate the Safety of COVID-19 Vaccination in Pregnant Women
Brief Title: Observational Maternal COVID-19 Vaccination Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Children's Hospital Medical Center, Cincinnati (Other); Boston Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107518
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2023-06

CONDITIONS: Pregnancy
Keywords: COVID-19 Vaccination; Immunizations in Pregnancy
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women who receive COVID-19 vaccine: Pregnant women who receive COVID-19 vaccine
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
This is a prospective, observational study. During the study, pregnant women will be followed post COVID-19 vaccination.

Injection-site (local) and systemic reaction data will be assessed on vaccination day and during the 7 days following the second vaccination using either identical web-based or paper diaries, depending on study participant preference.

Maternal serum samples will be collected for antibody titers relevant to COVID-19 at time points that include: prior to vaccination, ~29 days post second vaccination, and at delivery. At Duke University, maternal and infant cord blood will be collected at delivery and analyzed for the same antibody titers. At other clinical sites, these delivery samples will only be collected if feasible.

Pregnant women will be followed through 90 days postpartum. with comprehensive obstetric and neonatal outcomes obtained from medical record review.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women 18-45 years of age at the time of consent, inclusive
2. Intention of receiving or within 1 day of receiving the first dose or only dose of COVID-19 vaccine based on Advisory Committee on Immunization Practices (ACIP) and American College of Obstetricians and Gynecologists (ACOG) guidelines in response to the FDA Emergency Use Authorization (EUA) and in conjunction with federal and local vaccination campaign distribution plans
3. Willing to provide informed consent in a written or electronic format
4. Gestational age at time of consent < 34 weeks 0 days based on reconciliation of last menstrual period and ultrasound dating. Estimated due date (EDD) and Gestational Age (GA-EDD) will be based on reconciliation of "sure" first day of the last menstrual period (LMP) and earliest dating ultrasound. If the LMP is uncertain, then the earliest dating ultrasound will be used to determine EDD and GA. If the ultrasound derived-EDD is in agreement with sure-LMP derived EDD, then the LMP-derived EDD is used to determine GA. If the ultrasound derived EDD is not in agreement with the LMP-derived EDD, the ultrasound-derived EDD is used to determine GA.
5. Intention of being available for entire study period and complete all relevant study procedures, including follow-up phone calls and collection of delivery information.
6. English or Spanish literate

Exclusion Criteria:

1. Has immunosuppression as a result of an underlying illness or medications, such as antirejection/transplant regiments or immunomodulatory agents. Stable HIV disease is permitted per the following parameters:

   a. Confirmed stable HIV disease defined as document viral load <50 copies/mL and CD4 count >200 within 6 months before enrollment, and on stable antiretroviral therapy for at least 6 months
2. Has known hepatitis B (HBV) or hepatitis C (HBC). Stable HBV or HBC are permitted per the following parameters:

   1. If known HBV: confirmed inactive chronic HBV infection: HBsAg present for ≥6 months and HBeAg negative, anti-HBe positive; serum HBV DNA <2000 IU/mL; persistently normal ALT or AST levels; in those who had liver biopsy, findings that confirm absence of significant necroinflammation
   2. If known HCV: evidence of sustained virological response for ≥12 weeks after treatment or without evidence of HCV RNA viremia (undetectable HCV RNA)
3. Use of oral, parenteral, or high-dose inhaled glucocorticoids
4. Has an active neoplastic disease (excluding non-melanoma skin cancer), including those who used anti-cancer chemotherapy or radiation therapy during the current pregnancy
5. Signs or symptoms of active preterm labor, defined as regular uterine contractions with cervical change (dilation/effacement)
6. Known fetal congenital anomaly, e.g. genetic abnormality or major congenital malformation based on antenatal ultrasound
7. Anyone who is already enrolled or plans to enroll in a randomized clinical trial with any drug, vaccine or medical device. Co-enrollment in behavioral or other observational intervention studies are allowed at any time.
8. Any condition which, in the opinion of the investigators, may pose a health risk to the subject or interfere with the evaluation of the study objectives.
9. Anyone who is a relative of any research study personnel or is an employee supervised by study staff.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 350 adult pregnant women aged 18-45 years at < 34 weeks gestation who plan on receiving COVID-19 vaccination during the current pregnancy in accordance with the Advisory Committee on Immunization Practices (ACIP) and American College of Obstetricians & Gynecologists (ACOG) national recommendations.
Sampling Method: Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Adverse pregnancy outcomes in pregnant women vaccinated with COVID-19 vaccine | 12 months
  As measured by the proportion of women experiencing one of the following:
  Adverse birth outcome is a composite of occurrence of at least one of the following: preterm birth, spontaneous abortion, fetal death, or neonatal death.

SECONDARY OUTCOMES:
Preterm birth after COVID-19 vaccination | 12 months
  As measured by proportions of preterm birth after COVID-19 vaccination
Combined fetal and neonatal death after COVID-19 vaccination | 12 months
  As measured by proportions of combined fetal and neonatal death after COVID-19 vaccination
Spontaneous abortion after COVID-19 vaccination | 12 months
  As measured by proportions of spontaneous abortion after COVID-19 vaccination
Pregnant women with moderate/severe solicited reactogenicity events (local and systemic) within 7 days after COVID-19 vaccination | 7 days
  As measured by proportions of pregnant women with moderate/severe solicited reactogenicity events (local and systemic) within 7 days after COVID-19 vaccination
Women with ≥ 1 severe local and/or systemic reactogenicity event after COVID-19 vaccination | 3 months
  As measured by proportion of women with ≥ 1 severe local and/or systemic reactogenicity event after COVID-19 vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Geeta K Swamy, MD, Principal Investigator — Duke University; Karen R Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (4):
- United States (4):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT04826640/Prot_001.pdf
  • Informed Consent Form (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT04826640/ICF_002.pdf